CLINICAL TRIAL: NCT03435874
Title: A Phase Ib Age De-escalation Dose-escalation Randomised, Double-blind, Controlled Study of the Safety and Immunogenicity of ChAd63 RH5 and MVA RH5 Given Intramuscularly at 0 and 2-months in Healthy Adults, Children and Infants in Tanzania
Brief Title: Safety and Immunogenicity of ChAd63 RH5 and MVA RH5 in Adults, Young Children and Infants Living in Tanzania
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Ifakara Health Institute (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC070
Record Dates: First submitted 2018-01-08; First posted 2018-02-19 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-01

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: A Phase Ib age de-escalation dose-escalation randomised, double-blind, controlled study of the safety and immunogenicity of heterologous prime-boost with the candidate malaria vaccines ChAd63 RH5 and MVA RH5
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Group 1 Active (Experimental): n=6. Age 18-35 years. 5x10 10 vp ChAd63 RH5 at D0 and 2x10 8 pfu MVA RH5 at D56.
  Interventions: Biological: ChAd63 RH5; Biological: MVA RH5
- Group 1 Comparator (Placebo Comparator): n=3. Age 18-35 years. Rabies vaccine at D0 and D56.
  Interventions: Biological: Rabies Vaccine
- Group 2a Active (Experimental): n=6. Age 1-6 years. 1x10 10 vp ChAd63 RH5 at D0 and 1x10 8 pfu MVA RH5 D56.
  Interventions: Biological: ChAd63 RH5; Biological: MVA RH5
- Group 2a Comparator (Placebo Comparator): n=3. Age 1-6 years. Rabies vaccine at D0 and D56.
  Interventions: Biological: Rabies Vaccine
- Group 2b Active (Experimental): n=12. Age 1-6 years. 5x10 10 vp ChAd63 RH5 at D0 and 2x10 8 pfu MVA RH5 D56.
  Interventions: Biological: ChAd63 RH5; Biological: MVA RH5
- Group 2b Comparator (Placebo Comparator): n=6. Age 1-6 years. Rabies vaccine at D0 and D56.
  Interventions: Biological: Rabies Vaccine
- Group 3a Active (Experimental): n=6. Age 6-11 months. 1x10 10 vp ChAd63 RH5 at D0 and 1x10 8 pfu MVA RH5 D56.
  Interventions: Biological: ChAd63 RH5; Biological: MVA RH5
- Group 3a Comparator (Placebo Comparator): n=3. Age 6-11 months. Rabies vaccine at D0 and D56.
  Interventions: Biological: Rabies Vaccine
- Group 3b Active (Experimental): n=12. Age 6-11 months. 5x10 10 vp ChAd63 RH5 at D0 and 2x10 8 pfu MVA RH5 D56.
  Interventions: Biological: ChAd63 RH5; Biological: MVA RH5
- Group 3b Comparator (Placebo Comparator): n=6. Age 6-11 months. Rabies vaccine at D0 and D56.
  Interventions: Biological: Rabies Vaccine

INTERVENTIONS:
Biological: ChAd63 RH5 — Vaccine
  Arms: Group 1 Active; Group 2a Active; Group 2b Active; Group 3a Active; Group 3b Active
Biological: MVA RH5 — Vaccine
  Arms: Group 1 Active; Group 2a Active; Group 2b Active; Group 3a Active; Group 3b Active
Biological: Rabies Vaccine — Vaccine
  Arms: Group 1 Comparator; Group 2a Comparator; Group 2b Comparator; Group 3a Comparator; Group 3b Comparator

SUMMARY:
This is a dose-escalation, age de-escalation randomised double-blind controlled Phase Ib trial to assess the safety, tolerability and immunogenicity of ChAd63-RH5 administered with MVA-RH5 in a heterologous prime-boost regimen. Adults (18-35 years), young children (1-6 years) and infants (6-11 months) will be enrolled in the study. Safety data will be collected for each of the vaccination regimens. The humoral and cellular immune responses generated by each of these regimens will be assessed.

DETAILED DESCRIPTION:
* Experimental design: Phase Ib, double blind, age de-escalation dose-escalation, randomized (2:1 ratio), controlled trial.
* Healthy adults (18-35 years), young children (1-6 years) and infants (6-11 months) will be screened; those determined to be eligible, based on the inclusion and exclusion criteria, will be enrolled in the study.
* Route of administration of ChAd63-RH5 (day 0) and MVA-RH5 (2 months): both vaccines will be administered by the intramuscular route to the left deltoid.
* Each participant will be observed for at least 1 hour after vaccination to evaluate and treat any acute adverse events (AEs).
* There will be 7-day follow-up period for solicited AEs post-vaccination: Day 0, 2 and 7 evaluations will be carried out by the study clinician at the study centre and day 1, 3, 4, 5 and 6 evaluations will be carried out by a trained community health worker in the participant's home, after each vaccination.
* There will be a 28-day (day of vaccination and 28 subsequent days) follow-up after each vaccine dose for reporting unsolicited symptoms.
* Serious adverse events (SAEs) will be recorded throughout the study period. Prior to vaccination, any SAEs due directly to study procedures will be captured. All SAEs will be captured beginning with the administration of the priming dose of ChAd63 RH5 and ending 4 months after the booster dose with MVA RH5.
* Antibodies to RH5_FL will be determined at baseline and 14, 28, 56, 63, 84, 112, 140 and 168 days after ChAd63 RH5 in all participants.
* Cellular immune responses to RH5 will be evaluated at baseline and 14 (adults only), 28, 56, 63, 84 and 168 days after ChAd63 RH5 in all participants.
* The duration of involvement in the study from enrolment will be approximately 6 months. The vaccination phase of the study takes 9 weeks and the post-vaccination follow-up lasts for 4 months after the last dose.

ELIGIBILITY:
Inclusion Criteria:

Only participants who meet all the inclusion criteria will be enrolled into the trial;

* Group 1: Healthy male or female adults aged 18-35 years at the time of enrolment with signed consent.
* Group 1 (Female only participants): Must be non-pregnant (as demonstrated by a negative urine pregnancy test), and provide consent of their willingness to take Depo-Provera contraceptive during the study and safety follow-up period.
* Groups 2a & 2b: Healthy male or female young children aged 1-6 years at the time of enrolment with signed consent obtained from parents or guardians.
* Groups 3a & 3b: Healthy male or female infants aged 6-11 months at the time of enrolment with signed consent obtained from parents or guardians.
* Planned long-term (at least 9 months from the date of recruitment) or permanent residence in Bagamoyo town.
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or young children and infants with Z-score of weight-for-age within ±2SD.

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
* Clinically significant history of skin disorder (psoriasis, contact dermatitis etc.), allergy, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease and neurological illness as judged by the PI or other delegated individual.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* Weight for age z-scores below 2 standard deviations of normal for age.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, Kathon, neomycin, betapropiolactone.
* Any history of anaphylaxis in relation to vaccination.
* Clinically significant laboratory abnormality as judged by the PI or other delegated individual.
* Blood transfusion within one month of enrolment.
* History of vaccination with previous experimental malaria vaccines.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG).
* Any other finding which in the opinion of the PI or other delegated individual would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area.
* Positive malaria by blood smear at screening.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 6 Months to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Solicited symptoms after vaccination. | 7-day surveillance after each vaccination
  Frequency and severity (according to internationally recognised grading tables) of local and systemic solicited adverse events will be recorded for 7 days after each vaccination. For each, a causal relationship between the adverse event and IMP will be assigned.
Unsolicited symptoms after each vaccination. | 28-day surveillance after each vaccination.
  Frequency and severity (according to internationally recognised grading tables) of unsolicited adverse events will be recorded for 28 days after each vaccination. For each, a causal relationship between the adverse event and IMP will be assigned.
Serious adverse events during the study period. | Surveillance from first dose of vaccine to end of study (approximately 6 months from first vaccination).
  All serious adverse events from the first dose of IMP until the end of the study (approximately 6 months from first vaccination) will be recorded, causality assigned and reported to the Chief Investigator (as the Sponsor's representative) within 24 hours of the Investigator being aware of the suspected SAE. The Safety Monitoring Committee will be notified immediately by the PI if SAEs are deemed possibly, probably or definitely related to study interventions.

SECONDARY OUTCOMES:
Anti-RH5 antibody concentration by ELISA. | At baseline, and days 14 (adults only), 28, 56, 70, 84, 112, 140 and 168 after the first vaccination.
  Evaluation of the magnitude of antibody responses to PfRH5 in adults, children and infants residing in a malaria endemic country, as measured by ELISA
Growth inhibition activity of sera from vaccinees on a panel of P. falciparum parasites. | At baseline, and days 14 (adults only), 28, 56, 70, 84, 112, 140 and 168 after the first vaccination.
  Evaluation of the quality of antibody responses to RH5 in adults, children and infants residing in a malaria endemic country, as measured by an assay of growth inhibition activity on the vaccinees' sera
Avidity of anti-RH5 antibodies by ELISA and surface plasmon resonance (SPR) and/or other assays (to be defined). | At baseline, and days 14 (adults only), 28, 56, 70, 84, 112, 140 and 168 after the first vaccination.
  Evaluation of the longevity of antibody responses to PfRH5 in adults, children and infants residing in a malaria endemic country, as measured by ELISA, SPR +/- other assays
Cellular immune responses to the RH5 by ELISpot assay and/or Intracellular Cytokine Staining (ICS) and/or other assays to be defined. | At baseline, and days 14 (adults only), 28, 56, 70, 84, 112, 140 and 168 after the first vaccination.
  Evaluation of the magnitude and quality of cellular immune responses to PfRH5 in adults, children and infants residing in a malaria endemic country, by ELISpot assay and/or Intracellular Cytokine Staining (ICS) and/or other assays to be defined.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, Principal Investigator — University of Oxford
Locations (1):
- Ifakara Health Institute Clinical Trial Facility, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: No